CLINICAL TRIAL: NCT04168567
Title: A Protocol for a Prospective Study to Compare the Endometrial Microbiome in Patients With Body Mass Index Over 30 kg/m² Versus Under 25 kg/m².
Brief Title: The Impact of Body Mass Index on the Endometrial Microbiome in IVF Treatments. Tampere Infertility Microbiome Project (TIMP).
Status: Completed | Type: Observational
Sponsor: Tampere University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: R18068
Record Dates: First submitted 2019-09-19; First posted 2019-11-19 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Infertility, Female
Keywords: Microbiome; Microbiota; Obesity
MeSH Terms: conditions — Infertility, Female; Obesity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Obese patients: Patients with a BMI higher than 30kg/m² will be included in the first group.
  Interventions: Diagnostic Test: Microbiome analysis
- Normal-weight patients: Patients with a BMI under 25 kg/m² will be included in the second group.
  Interventions: Diagnostic Test: Microbiome analysis

INTERVENTIONS:
Diagnostic Test: Microbiome analysis — Samples from TIMP microbiome project will be analyzed with NGS techniques.

SUMMARY:
This study project is an observational trial involving 90 patients suffering from male type infertility. The patients are divided in two groups (45 patients per group) based on their body mass index (BMI).

DETAILED DESCRIPTION:
This study (Tampere Infertility Microbiome Project, TIMP) aims to clarify the differences in the microbiome variety between obese and normal-weight patients. The first group will consist of patients with the body mass index (BMI) over 30 kg/m², while the second group will include patients with a healthy weight BMI under 25. The samples will be collected at the time of embryo transfer and analyzed in a laboratory specialing in next-generation sequencing (NGS) techniques.

ELIGIBILITY:
Inclusion Criteria:

* Patients with male infertility scheduled for IVF treatment and fresh embryo transfer
* Primary or secondary male-type infertility
* BMI over 30 kg/m² or under 25 kg/m²
* Patient's willingness to participate

Exclusion Criteria:

* Patients with endometriosis or adenomyosis
* Use of antibiotics during IVF treatment or oocyte retrieval
* Technical diffuculties in embryo transfer or no embryos available for transfer

Ages: 20 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Obese and non-obese female with male-infertility
Sampling Method: Non-Probability Sample
Enrollment: 91 (Actual)
Dates: Start 2020-08-14 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Microbiome variety between groups | through study completion, 1-2 years from the starting date
  This study aims to investigate differences of endometrium microbiome and continuum of microbiota from anal to reproductive tract site between obese and normal-weight patients. Samples will be collected at the time of embryo transfer using embryo transfer catheter. The study will also examine pregnancy outcomes and microbiome differences in pregnant patients.

SECONDARY OUTCOMES:
Ongoing pregnancy rate | up to 2-3 months
  Ongoing pregnancy rate

CONTACTS AND LOCATIONS:
Overall Officials: Katja Ahinko, Principal Investigator — Tampere University Hospital
Locations (1):
- Tampere University Hospital, Tampere, Finland